CLINICAL TRIAL: NCT00853450
Title: A Randomised, Open-label, Single-Centre, Phase I, Crossover Study to Evaluate the Effect of AZD6482, Compared With Clopidogrel, on Bleeding Time in Healthy Volunteers Receiving Low-Dose ASA
Brief Title: Bleeding Time Study With AZD6482, Clopidogrel and ASA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Peter Held, Medical Science Director, Early Thrombosis & Haemostasis, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1700C00004; EudraCT no. 2008-007030-21
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Antiplatelet Effect
Keywords: Antiplatelet
MeSH Terms: interventions — 2-(1-(7-methyl-2-morpholin-4-yl-4-oxo-4H-pyrido(1,2-a)pyrimidin-9-yl)ethylamino)benzoic acid; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD6482 on top of ASA
  Interventions: Drug: AZD6482; Drug: ASA
- 2 (Active Comparator): Clopidogrel on top of ASA
  Interventions: Drug: Clopidogrel; Drug: ASA

INTERVENTIONS:
Drug: AZD6482 — Single intravenous infusion during a maximum of 5 hours
  Arms: 1
Drug: Clopidogrel — Oral doses given once daily during 7 days. 300 mg on day 1 and 75 mg on day 2 to 7.
  Other Names: Plavix®
  Arms: 2
Drug: ASA — 75 mg orally once daily during 7 days in each treatment arm
  Other Names: Trombyl®

SUMMARY:
The primary purpose of this study is to evaluate the effect of AZD6482 and clopidogrel on bleeding time when taken together with low-dose ASA.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19.0 and 30.0 kg/m2, inclusive and body weight between 50.0 and 100.0 kg, inclusive
* Provision of written informed consent

Exclusion Criteria:

* Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms.
* Acute illness, surgical procedure or trauma from 2 weeks before pre-entry visit until the first baseline visit or clinically significant abnormalities in clinical chemistry, haematology, urinalysis or supine BP or pulse
* Known impaired glucose tolerance, known galactose intolerance, total lactase deficiency or glucose-galactose malabsorption or known or suspected Gilbert's syndrome

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-02; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Capillary Bleeding Time (CBT) | Prior to first dose in each treatment period, on study day 6 and 7 in treatment period A and on study day 7 in treatment period B

SECONDARY OUTCOMES:
Effect on bleeding | Prior to first dose in each treatment period, twice on study day 6 and three times on study day 7 in treatment period A and twice on study day 7 in treatment period B
Pharmacokinetics | Prior to AZD6482 infusion and repeatedly during 6 hours after end of infusion
Safety variables (adverse events, blood pressure, pulse, ECG, safety lab) | Repeatedly during the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Held, Study Director — AstraZeneca Mölndal; Bo Fransson, MD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Lund
Locations (1):
- Research Site, Lund, Sweden